CLINICAL TRIAL: NCT03087279
Title: A Cluster Randomized Control Trial to Assess the Impact of Active Learning on Child Activity, Attention Control, and Academic Outcomes: The Texas I-CAN Trial
Brief Title: Assessing Impact of Active Learning on Student Outcomes: Texas Initiatives for Children's Activity and Nutrition (ICAN)
Acronym: ICAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1R01HD070741 (NIH)
Record Dates: First submitted 2017-03-09; First posted 2017-03-22 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Texas I-CAN Active Math Lessons (Experimental): Texas I-CAN Active math lesson in academic classroom
  Interventions: Behavioral: Texas I-CAN!
- Texas I-CAN Active Language Arts Lessons (Experimental): Texas I-CAN Active language arts lessons in academic classroom
  Interventions: Behavioral: Texas I-CAN!
- Control (No Intervention): Regular, Sedentary academic lessons in math and language arts

INTERVENTIONS:
Behavioral: Texas I-CAN! — physically active, academic lessons in the elementary school classroom
  Arms: Texas I-CAN Active Language Arts Lessons; Texas I-CAN Active Math Lessons

SUMMARY:
Background: Active learning is designed to pair physical activity with the teaching of academic content. This has been shown to be a successful strategy to increase physical activity and improve academic performance. The existing designs have confounded academic lessons with physical activity. As a result, it is impossible to determine if the subsequent improvement in academic performance is due to: (1) physical activity, (2) the academic content of the active learning, or (3) the combination of academic material taught through physical activity.

Methods / Design: The Texas I-CAN project is a 3-arm, cluster randomized control trial in which 28 elementary schools were assigned to either control, math intervention, or spelling intervention. As a result, each intervention condition serves as an unrelated content control for the other arm of the trial, allowing the impact of physical activity to be separated from the content. That is, schools that perform only active math lessons provide a content control for the spelling schools on spelling outcomes. This also calculated direct observations of attention and behavior control following periods of active learning.

Discussion: This design is unique in its ability to separate the impact of physical activity, in general, from the combination of physical activity and specific academic content. This, in combination with the ability to examine both proximal and distal outcomes along with measures of time on task will do much to guide the design of future, school-based interventions.

ELIGIBILITY:
Inclusion Criteria:

* students in 4th grade in a participating elementary school and their 4th grade teachers

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2716 (Actual)
Dates: Start 2012-08-15 (Actual); Primary Completion 2015-05-31 (Actual); Study Completion 2015-05-31 (Actual)

PRIMARY OUTCOMES:
Physical activity level | one school week
  time in moderate to vigorous physical activity
Time on task | change in time on task from baseline to 15 minutes post academic lesson
  student attentional focus in the classroom 15 minutes prior to and 15 minutes post active lesson implemented in the classroom on one school day
Acute academic achievement | change in math and language arts scores from Baseline to 2 weeks
  acute academic scores on math and language arts test developed by fourth grade teacher
Long-term math achievement | Change in math achievement scores from Baseline to 7 months
  Academic scores on math sub tests (Calculation, Fluency) of the Woodcock Johnson III
Long-term language arts achievement | Change in language arts achievement from Baseline to 7 months
  Academic scores on spelling sub test of the Woodcock Johnson III and comprehension section of Gates MacGinitie test

CONTACTS AND LOCATIONS:
Overall Officials: John B Bartholomew, PHD, Principal Investigator — UT Austin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bartholomew JB, Jowers EM, Errisuriz VL, Vaughn S, Roberts G. A cluster randomized control trial to assess the impact of active learning on child activity, attention control, and academic outcomes: The Texas I-CAN trial. Contemp Clin Trials. 2017 Oct;61:81-86. doi: 10.1016/j.cct.2017.07.023. Epub 2017 Jul 22. PMID 28739542